CLINICAL TRIAL: NCT04282369
Title: Evaluation Of The Efficacy Of Four Different Non-invasive Ventilation Modes Performed In The Delivery Room In Late Preterm And Term Infants Wıth Respiratory Distress
Brief Title: Evaluation Of The Efficacy Of Four Different Non-invasive Ventilation Modes Performed In The Delivery Room
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ilker Gönen, Neonatologist, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 32342545
Record Dates: First submitted 2020-02-17; First posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Respiratory Disease; Respiratory Insufficiency
Keywords: respiratory distress, newborn, noninvasive ventilation
MeSH Terms: conditions — Respiration Disorders; Respiratory Insufficiency; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HHFNC (Active Comparator): In this group patients will receive respiratory support by high flow nasal cannula.
  Interventions: Device: HHHFNC
- nCPAP (Active Comparator): In this group patients will receive respiratory support by nasal CPAP.
  Interventions: Device: NCPAP
- nIPPV (Active Comparator): In this group patients will receive respiratory support by nasal IPPV.
  Interventions: Device: NIPPV
- nHFO (Active Comparator): In this group patients will receive respiratory support by nasal high frequency oscillatory. ventilation.
  Interventions: Device: NHFO

INTERVENTIONS:
Device: HHHFNC — noninvasive ventilation modality
  Arms: HHFNC
Device: NCPAP — noninvasive ventilation modality
  Arms: nCPAP
Device: NIPPV — noninvasive ventilation modality
  Arms: nIPPV
Device: NHFO — noninvasive ventilation modality
  Arms: nHFO

SUMMARY:
Evaluation Of The Efficacy Of Four Different Non-invasive Ventilation Modes Performed In The Delivery Room In Late Preterm And Term Infants Wıth Respiratory Distress

DETAILED DESCRIPTION:
In this study, it is aimed to search the efficacy and comfort of the four different non-invasive ventilation modes in the delivery room. HHFNC, NCPAP, NIPPV and NHFO modes are used for the respiratory distress of the late preterm and term babies.

ELIGIBILITY:
Inclusion Criteria:

* late preterm and term infants with respiratory distress

Exclusion Criteria:

* intubation for the respiratory distres.
* major abnormalities

Max Age: 2 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2020-02-18 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
Silverman Score | 6 months
  The respiratory status of the newborns will be evaluated with the scoring system defined by Silverman.

SECONDARY OUTCOMES:
N-PASS score | 6 months
  evaluation of the comfort of the four different noninvasive ventilation modes

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Suleyman Research and Training Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No